CLINICAL TRIAL: NCT04603365
Title: A Phase 2 Study of Pamiparib (BGB-290) Plus Temozolomide for Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC)
Brief Title: Pamiparib and Temozolomide for the Treatment of Hereditary Leiomyomatosis and Renal Cell Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: BeiGene (Industry); Driven To Cure (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001106; NCI-2020-05351 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-10

CONDITIONS: Clear Cell Papillary Renal Neoplasm; Collecting Duct Carcinoma; Hereditary Leiomyomatosis and Renal Cell Carcinoma; Hereditary Papillary Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Unclassified Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Stage III Renal Cell Cancer American Joint Committee on Cancer (AJCC) v8; Stage IV Renal Cell Cancer AJCC v8; Tubulocystic Renal Cell Carcinoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Hereditary leiomyomatosis and renal cell cancer | interventions — pamiparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pamiparib, temozolomide) (Experimental): Patients receive PO BID on days 1-28 and temozolomide PO QD on days 1-7. Cycles repeat every 28 days for up to 36 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pamiparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Pamiparib — Given PO
  Other Names: BGB-290; PARP Inhibitor BGB-290
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial investigates how well pamiparib and temozolomide work in treating patients with hereditary leiomyomatosis and renal cell (kidney) cancer. Poly adenosine diphosphate-ribose polymerase (PARPs) are proteins that help repair DNA mutations. PARP inhibitors, such as pamiparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pamiparib and temozolomide may help treat patients with hereditary leiomyomatosis and renal cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate response rate of pamiparib plus low-dose temozolomide.

SECONDARY OBJECTIVES:

I. To evaluate the progression-free survival with pamiparib plus low-dose temozolomide.

II. To evaluate the safety (adverse events [AE's]) with pamiparib plus low-dose temozolomide.

TRANSLATIONAL OBJECTIVES:

I. To determine the association between plasma and tumor 2-hydroxyglutarate (2HG), fumarate, and succinate levels and response to treatment.

II. To analyze the association of the genomic mutational signature (by whole genome sequencing) of the tumor to treatment.

OUTLINE:

Patients receive orally (PO) twice daily (BID) on days 1-28 and temozolomide PO once daily (QD) on days 1-7. Cycles repeat every 28 days for up to 36 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily agreed to participate by signing an informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Ability to swallow whole capsules
* Histologically confirmed metastatic or unresectable renal cell carcinoma with morphologic features consistent with hereditary leiomyomatosis and renal cell cancer (HLRCC). This can include tumors with overlapping morphology previously called papillary, tubulocystic, tubulopapillary, collecting duct, or unclassified as long as in the HLRCC- spectrum
* The presence of a documented germline fumarate hydratase (FH) alteration (mutation or deletion). This includes pathogenic or likely pathogenic alterations but may also include variants of unknown significance (VUS) in patients with strong personal or family history where the clinician makes a presumed clinical diagnosis
* Progression on 1 or more lines of systemic therapies for metastatic disease. Neo/adjuvant therapy in the absence of documented distant disease does not count as a line of therapy
* No known intolerance of study drugs or excipients, and able to comply with study requirements
* Absolute neutrophil count (ANC) >= 1,500 /microliter (mcL) (< 2 weeks prior to day 1)
* Platelets >= 100,000 / mcL (< 2 weeks prior to day 1)
* Hemoglobin >= 10 g/dL or >= 6.2 mmol/L without transfusion or erythropoietin (EPO) dependency (within 2 weeks of first dose)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 40 mL/min for participants with creatinine levels > 1.5 x institutional ULN (< 2 weeks prior to day 1)

  * Creatinine clearance should be calculated using the standard Cockcroft and Gault equation
* Total serum bilirubin =< 1.5 x ULN (total bilirubin must be < 4 x ULN for subject with Gilbert's syndrome) (< 2 weeks prior to day 1)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN OR =< 5 x ULN for participants with liver metastases (< 2 weeks prior to day 1)
* International normalized ratio (INR) or prothrombin time (PT), and activated partial thromboplastin time (aPTT) =<1.5 x ULN unless participant is receiving anticoagulant therapy, and then only as long as PT or PTT is within therapeutic range of intended use of anticoagulants (< 2 weeks prior to day 1)
* Female patients of childbearing potential and female partners of male study patients must agree to practice highly effective methods of birth control for the duration of the study and for >= 6 months after the last dose of study drug. In addition, non-sterile male patients must agree to practice highly effective methods of birth control and avoid sperm donation for the duration of the study and for >= 6 months after the last dose of study drug
* From the time of the first study-drug treatment through 180 days after the last study drug treatment, male participants must use a condom when 1) having sex with a pregnant woman AND 2) having sex with a woman of childbearing potential
* Male and female participants must agree not to donate sperm or eggs, respectively, from the first study-drug treatment through 180 days after the last study drug treatment
* Female participants must agree to not breastfeed during the study or for 180 days after the last dose of study treatment
* If available, agreement to provide archival tumor tissue for exploratory biomarker analyses
* Willingness to undergo a fresh tumor biopsy if deemed safe and feasible by the investigator

Exclusion Criteria:

* Known hypersensitivity to any temozolomide (TMZ) component
* Prior treatment with a PARP inhibitor
* Received chemotherapy, biologic therapy, immunotherapy, or investigational agent within 3 weeks (or =< 5 half-lives, whichever is shorter) prior to cycle 1/day 1
* Have any unresolved acute effects of any prior therapy of grade 2 or higher, except for AEs not constituting a safety risk by investigator judgment
* Had a major surgical procedure (per investigator discretion) =< 4 weeks prior to cycle 1/day 1, or anticipation of need for major surgical procedure during the course of the study
* Have other diagnosis of malignancy

  * Except for surgically excised non-melanoma skin cancer, adequately treated carcinoma in situ of the cervix, localized prostate cancer treated with curative intent, adequately treated low-stage bladder cancer, ductal carcinoma in situ treated surgically with curative intent, or a malignancy diagnosed > 2 years ago, with no current evidence of disease and no therapy =< 2 years prior to day 1
* Subject who has received local radiotherapy of non-target lesions for local symptom control within the last 4 weeks must have recovered from any adverse effects of radiotherapy before recording baseline symptoms
* Have untreated leptomeningeal or brain metastasis. Subject with previously treated brain metastases is eligible if the metastases have shown no progression on brain computed tomography (CT) or magnetic resonance imaging (MRI) over at least 4 weeks, the subject has no symptoms due to the brain metastases, and the subject has been off corticosteroids for >= 2 weeks
* Have active infection requiring systemic treatment
* Have known human immunodeficiency virus (HIV) infection
* No known chronic active liver disease or evidence of acute or chronic hepatitis B virus (HBV) or hepatitis C (HCV) infection. Patients with prior curative treatment of hepatitis C virus are allowed if treated > 2 weeks prior to treatment previously and HCV ribonucleic acid (RNA) undetectable by established laboratory values
* Have any of the following cardiovascular criteria:

  * Current evidence of cardiac ischemia
  * Current symptomatic pulmonary embolism
  * Acute myocardial infarction =< 6 months prior to cycle 1/ day 1
  * Heart failure of New York Heart Association classification III or IV =< 6 months prior to cycle 1/ day 1
  * Grade >= 2 ventricular arrhythmia =< 6 months prior to cycle 1/ day 1
  * Cerebral vascular accident (CVA) =< 6 months prior to cycle 1/ day 1
* Have an active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease or had previous complete gastric resection or lap band surgery

  * Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed (assuming no drug interaction potential)
* Use or have anticipated need for food or drugs known to be strong or moderate cytochrome P450 (CYP)3A inhibitors or strong CYP3A inducers =< 10 days (or =< 5 half-lives, whichever is shorter) prior to day 1
* Are pregnant or nursing (females of childbearing potential require a negative serum pregnancy test =< 7 days before day 1)
* Requirement for intravenous (IV) alimentation (at the time of randomization)
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participants must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-05-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 36 months of treatment
  Defined as total number of subjects with confirmed responses of either complete response (CR) or partial response (PR) divided by the total number of subjects in the response-evaluable population per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 by investigator assessment. Response rate will be calculated along with the corresponding exact one-sided 95% Clopper-Pearson confidence interval.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the first dose of study drug to the date of progressive disease first documented disease progression per RECIST v1.1 or death due to any cause by investigator assessment, whichever occurs first, assessed up to 3 years after completion of treatment
  PFS will be summarized using the Kaplan Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.
Incidence of adverse events (AEs) | Up to 36 months
  Safety profile including AE and serious (S)AEs will be reported. Simple descriptive statistics will be used to summarize toxicities in terms of type, severity (by Common Terminology Criteria for Adverse Events [CTCAE] v4.03 toxicity table) and minimum or maximum values for laboratory measures, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects. Adverse events will be tabulated and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.

OTHER OUTCOMES:
Plasma and tumor 2-hydroxyglutarate (2HG), fumarate, and succinate levels | Up to 36 months
  Plasma and tumor samples will be subjected to multiplex liquid chromatography coupled with tandem mass spectrometry. Will determine the association between plasma and tumor 2HG, fumarate, and succinate levels and response to treatment.
Genomic mutational signature (by whole genome sequencing) | Up to 36 months
  Tumor material will be subjected to whole genome sequencing to determine the mutational spectrum. Will analyze the association of the genomic mutational signature of the tumor to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shuch, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center